CLINICAL TRIAL: NCT05551182
Title: The Study of Efficacy on Low Dose Nicergoline in Dysphagia Patients Compares With High Dose Nicergoline.
Brief Title: Nicergoline Use in Dysphagia Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Collaborators: Silpakorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDY-2022
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Dysphagia
Keywords: Dysphagia; Stroke; Parkinson's disease; Dementia; Dysphagia improvement; Nicergoline
MeSH Terms: conditions — Deglutition Disorders; Stroke; Parkinson Disease; Dementia | interventions — Nicergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicergoline low dose (Experimental): Nicergoline 10 mg bid (20 mg/day)
  Interventions: Drug: Nicergoline
- Nicergoline high dose (Experimental): Nicergoline 30 mg bid (60 mg/day)
  Interventions: Drug: Nicergoline

INTERVENTIONS:
Drug: Nicergoline — The participants in both arms will receive nicergoline for treatment dysphagia 12 weeks.
  Other Names: Sermion

SUMMARY:
Dysphagia is a complication in patient with stroke, Parkinson's disease or dementia that can lead to aspiration pneumonia. This study aimed to investigate dysphagia improvement after treatment with nicergoline low dose and high dose, the relationship between nicergoline dose and clinical improvements, side effect of nicergoline and simulation optimal nicergoline dose in dysphagia improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 20 years
* Stroke (post events at least 2 months), Parkinson's disease and dementia patients who have dysphagia symptom
* Do not take nicergoline prior recruit 2 weeks
* Continue current medications
* Consent to join

Exclusion Criteria:

* Allergy to gentamicin or components
* On anticoagulants including Heparin, Enoxaparin, Fondaparinux, Warfarin, Dabigatran, Apixaban, Rivaroxaban and Edoxaban
* On antiplatelet > 1 drug (ex. dual antiplatelet)
* On ACE-I or Dopaminergic agent 2 months or less
* Chronic dyspepsia
* Chronic gout or hyperuricemia > 8 mg/dL
* CrCl < 30 ml/min
* Impair hepatic function including child puge B, C or active hepatitis
* Brainstem stroke
* Parkinson plus syndrome: PSP, MSA, DLB, etc
* Advanced cancer or other medical conditions
* Bed ridden
* Laryngopharynx surgery
* SBP<100 or DBP 60 mmHg
* HR<50/min
* Active bleeding
* Pregnancy or lactation
* Known of poor compliance for any treatments

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Rate of dysphagia improvement in low dose nicergoline compare with high dose nicergoline group. | 4 and 12 weeks
  Dysphagia improvement evaluated by physician with GUSS method after nicergoline administration in 4 and 12 week.
Rate of dysphagia improvement in low dose nicergoline and high dose nicergoline group compare pre and post nicergoline treatment each group. | 4 and 12 weeks
  Dysphagia improvement evaluated by physician with GUSS method after nicergoline administration in 4 and 12 week.
Relation between MDL level, substanceP and dysphagia improvement after nicergoline administration both groups (low dose and high dose) in steady state. | 4 weeks
  Blood sampling for MDL level in Ctrough, Cpeak and substanceP at steady state of nicergoline effect.

SECONDARY OUTCOMES:
Optimal nicergoline dose for dysphagia improvement. | 12 weeks
  Simulated optimal nicergoline dose by Monte Carlo method with Ctrough, Cpeak and dysphagia improvement
Incidence of aspiration pneumonia in low dose nicergoline compare with high dose nicergoline group. | 12 weeks
  Evaluated by clinical reported from patients and hospitalization data.
Rate of cognitive function improvement in low dose nicergoline compare with high dose nicergoline group. | 12 weeks
  Evaluated by physician with MMSE-Thai 2002 after nicergoline administration in 12 weeks.
Rate of cognitive function improvement in low dose nicergoline and high dose nicergoline group compare pre and post nicergoline treatment each group. | 12 weeks
  Evaluated by physician with MMSE-Thai 2002 after nicergoline administration in 12 weeks.
Adverse side effect in low dose and high dose nicergoline treatment. | 4 and 12 weeks
  Blood sampling for renal function (including creatinine serum, creatinine clearance) and uric serum. Other adverse side effect reported by patients/care givers.

CONTACTS AND LOCATIONS:
Overall Officials: Jutikan Imsub, PharmD, Study Chair — College of Pharmacy, Burapha university; Sittichoke Sirimontakan, MD, Principal Investigator — Phramongkutklao hospital and College of Medicine; Juthathip Suphanklang, BCP, Study Director — Phramongkutklao hospital and College of Medicine; Pasiri Sithinamsuwan, MD, Study Director — Phramongkutklao hospital and College of Medicine
Locations (1):
- Phramongkutklao Hospital, Ratchathewi, Bangkok, Thailand